CLINICAL TRIAL: NCT01771809
Title: A Multicenter Open-Label Extension Study To Assess Long-Term Safety Of PF-00547659 In Subjects With Ulcerative Colitis (TURANDOT II)
Brief Title: Long-Term Safety Of PF-00547659 In Ulcerative Colitis
Acronym: TURANDOT II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A7281010; 2012-002031-28 (EudraCT Number); TURANDOT II (Other: Alias Study Number)
Record Dates: First submitted 2013-01-08; First posted 2013-01-18 (Estimated); Results first posted 2019-04-18 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Ulcerative Colitis
Keywords: Anti-TNF Refractory; Active Ulcerative Colitis; Immunosuppressant Refractory
MeSH Terms: conditions — Colitis, Ulcerative | interventions — ontamalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SHP647 75 mg (Experimental): Participants will receive 75 milligrams (mg) of SHP647 subcutaneous (SC) injection every 4 weeks for 72 weeks in the anterolateral right/left thigh or the deltoid area or the abdomen. During the first 72 weeks, a one time dose escalation to 225 mg of SHP647 SC injection every 4 weeks is allowed after 8 weeks of the study for participants who experience clinical deterioration or unacceptably low level of response to the investigational product. The decision to escalate will be guided by the response and relapse criteria tempered by clinical judgment. Following the first 72 weeks, participants will receive 75 mg of SHP647 SC injection every 4 weeks for an additional 72 weeks in the anterolateral right/left thigh or the deltoid area or the abdomen.
  Interventions: Drug: 75mg SHP647 (PF-00547659)
- SHP647 225 mg (Experimental): Participants will receive 225 mg of SHP647 SC injection every 4 weeks for 72 weeks followed by 75 mg of SHP647 SC injection every 4 weeks for an additional 72 weeks in the anterolateral right/left thigh or the deltoid area or the abdomen.
  Interventions: Drug: 225mg SHP647 (PF-00547659)

INTERVENTIONS:
Drug: 75mg SHP647 (PF-00547659) — 75 mg sterile liquid injected subcutaneously every 4 weeks.
  Arms: SHP647 75 mg
Drug: 225mg SHP647 (PF-00547659) — 225 mg sterile liquid injected subcutaneously every 4 weeks.
  Arms: SHP647 225 mg

SUMMARY:
Subjects with Ulcerative Colitis who have completed an induction study with PF-00547659 will receive an additional 144 weeks of open-label treatment to evaluate the long-term safety of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 18 and 66 years of age.
* Subjects previously enrolled in study A7281009 (NCT01620255) who have completed the 84 day (12 week) induction period.

Exclusion Criteria:

* Subjects that have completed Day 84 (Week 12) of study A7281009 but have experienced serious event(s) related to the investigational product, an unstable medical condition, or any other reason, in the opinion of the investigator, would preclude entry or participation in this study.
* Subjects who are taking any dose of Azathioprine (AZA), 6-mercaptopurine(6 MP) or Methotrexate (MTX).

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2013-03-18 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2017-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shire Director, Study Director — Takeda
Locations (99):
- United States (29):
  - Mayo Clinic Arizona - Scottsdale, Scottsdale, Arizona
  - UCSD Altman Clinical and Translational Research Institute, La Jolla, California
  - Community Clinical Trials, Orange, California
  - Rocky Mountain Gastroenterology, Thornton, Colorado
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - Nature Coast Clinical Research, Inverness, Florida
  - Bassan and Bloom M.D.s, Miramar, Florida
  - Internal Medicine Specialists, Orlando, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Atlanta Gastroenterology Specialists, PC, Suwanee, Georgia
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Commonwealth Clinical Studies, Brockton, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Minnesota Gastroenterology, PA, Plymouth, Minnesota
  - Center for Digestive and Liver Diseases, Mexico, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nevada School of Medicine, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Albany Medical College, Albany, New York
  - Weill Cornell Medical College of Cornell University, New York, New York
  - Premier Medical Group of the Hudson Valley, PC, Poughkeepsie, New York
  - UNC Memorial Hospital, Chapel Hill, North Carolina
  - The Oregon Clinic-West Hills Gastroenterology Associates, P.C., Portland, Oregon
  - Gastro One, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College Of Medicine - Baylor Medical Center, Houston, Texas
  - McGuire DVAMC, Richmond, Virginia
  - Univeristy of Washington, Seattle, Washington
  - Allegiance Research Specialists, Wauwatosa, Wisconsin
- Australia (6):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Mater Health Services, South Brisbane, Queensland
  - Alfred Hospital, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
- AKH Wien, Universitaetsklinik fuer Innere Medizin III, Vienna, Austria
- Belgium (3):
  - AZ St. Elisabeth Herentals, Herentals
  - University Hospital Gasthuisberg, Leuven
  - Centre Hospitalier de Mouscron, Mouscron
- MBAL Sveti Ivan Rilski, Klinika po Gastroenterologia, Sofia, Bulgaria
- Canada (7):
  - (G.I.R.I.) GI Research Institute, Vancouver, British Columbia
  - Percuro Clinical Research, Ltd, Victoria, British Columbia
  - Hamilton Health Sciences Corp, McMaster Univ Medical Centre, Hamilton, Ontario
  - London Health Sciences Centre - University Hospital, London, Ontario
  - Taunton Surgical Centre, Oshawa, Ontario
  - Universite de Montreal - Hopital Maisonneuve-Rosemont (HMR), Montreal, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
- Czechia (3):
  - Hepato-Gastroenterologie HK s.r.o. Poliklinika III, Hradec Králové
  - IBD Clinical and Research Centre, Prague
  - Krajska zdravotni, a.s., Masarykova nemocnice v Usti nad Labem, Ústí nad Labem
- France (6):
  - CHU Amiens-Picardie - Hopital Sud, Amiens
  - Centre Hospitalier Universitaire (CHU) de Caen - Hopital Cote de Nacre, Caen
  - Hopital Huriez CHRU de Lille, Lille
  - CHU De Nice Hopital De L'Archet II, Nice
  - CHU de Saint-Etienne Hopital Nord, Saint-Priest-en-Jarez
  - CHU de Nancy - Hopital Brabois, Vandœuvre-lès-Nancy
- Germany (2):
  - Universitaetsklinikum Schleswig-Holstein, Campus Kiel, Kiel, Schleswig-Holstein
  - Universitaetsklinikum Regensburg, Klinik und Poliklinik fuer Innere Medizin 1, Regensburg
- Csongrad Megyei Dr. Bugyi Istvan Korhaz, Szentes, Csongrád megye, Hungary
- Israel (4):
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Ein Kerem University Hospital - Gastroenterology and Liver Diseases Unit, Jerusalem
  - Meir Medical Center, Kfar Saba
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Italy (7):
  - Universita' degli Studi "Magna Graecia" di Catanzaro, Catanzaro
  - Milan University, Humanitas Clinical Institute, Milan
  - Policlinico Universitario Campus Bio-Medico, Roma
  - Azienda Ospedaliera Universitaria, Policlinico Tor Vergata, Roma
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - Universita Cattolica del Sacro Cuore, Roma
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
- Netherlands (3):
  - Academic Medical Center, Amsterdam
  - University Medical Center Groningen (UMCG), Groningen
  - Maastricht University Medical Center, Maastricht
- New Zealand (2):
  - Christchurch Hospital, Christchurch, Canterbury
  - Waikato Hospital, Hamilton
- Poland (7):
  - Centrum Endoskopii Zabiegowej, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Centrum Medyczne-Szpital Swietej Rodziny Sp.z.o.o., Lodz, Wojlodzkie
  - Gabinet Endoskopii Przewodu Pokarmowego, Krakow
  - NZOZ Centrum Medyczne HCP sp. z o.o, Poznan
  - Klinika Chorob Wewnetrznych I Gastroenterologii, Warsaw
  - Niepubliczny Zaklad Opieki Zdrowotnej VIVAMED, Warsaw
  - Lexmedica, Wroclaw
- St. Petersburg State Medical Academy for Postgraduate Education, Saint Petersburg, Russia
- Serbia (3):
  - Military Medical Academy, Belgrade
  - Clinical Hospital Center Zemun, Belgrade
  - Clinical Hospital Centre Bezanijska Kosa, Belgrade
- Slovakia (3):
  - Ustredna vojenska nemocnica SNP Ruzomberok - Fakultna nemocnica, Nitra
  - Gastro L., s.r.o., Prešov
  - Ustredna vojenska nemocnice SNP Ruzomberok - Fakultna nemocnica, Ružomberok
- Kingsbury Hospital, Claremont, Cape Town, South Africa
- South Korea (5):
  - Yeungnam University Medical Center, Daegu
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (4):
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Centro Medico Teknon-Institut de la Macula i de la Retina, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Parc de Salut Mar-Hospital del Mar, Barcelona

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7281010&StudyName=Long-Term%20Safety%20Of%20PF-00547659%20In%20Ulcerative%20Colitis

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 101 centers in 21 countries between 18 Mar 2013 (first participant first visit) and 13 Dec 2017 (last participant last visit).
Pre-assignment Details: A total of 331 participants were randomized and 330 participants received treatment in the study. One participant discontinued due to adverse event prior to receiving treatment.
Groups:
- SHP647 75 mg: Participants received 75 milligrams (mg) of SHP647 subcutaneous (SC) injection every 4 weeks for 72 weeks in the anterolateral right/left thigh or the deltoid area or the abdomen. During the first 72 weeks, a one time dose escalation to 225 mg of SHP647 SC injection every 4 weeks was allowed after 8 weeks of the study for participants who experienced clinical deterioration or unacceptably low level of response to the investigational product. The decision to escalate was guided by the response and relapse criteria tempered by clinical judgment. Following the first 72 weeks, participants received 75 mg of SHP647 SC injection every 4 weeks for an additional 72 weeks in the anterolateral right/left thigh or the deltoid area or the abdomen.
- SHP647 225 mg: Participants received 225 mg of SHP647 SC injection every 4 weeks for 72 weeks followed by 75 mg of SHP647 SC injection every 4 weeks for an additional 72 weeks in the anterolateral right/left thigh or the deltoid area or the abdomen.
Period: Overall Study
Arm/Group | SHP647 75 mg | SHP647 225 mg
Started | 164 | 166
Completed | 93 | 83
Not Completed | 71 | 83
Not completed — Adverse Event | 4 | 12
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 34 | 42
Not completed — Lost to Follow-up | 1 | 3
Not completed — Other (Insufficient clinical response) | 22 | 20
Not completed — Death | 1 | 0
Not completed — Other (other) | 9 | 5

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAS) consisted of all enrolled participants who had received at least 1 dose of SHP647.
Groups:
- SHP647 75 mg: Participants received 75 mg of SHP647 SC injection every 4 weeks for 72 weeks in the anterolateral right/left thigh or the deltoid area or the abdomen. During the first 72 weeks, a one time dose escalation to 225 mg of SHP647 SC injection every 4 weeks was allowed after 8 weeks of the study for participants who experienced clinical deterioration or unacceptably low level of response to the investigational product. The decision to escalate was guided by the response and relapse criteria tempered by clinical judgment. Following the first 72 weeks, participants received 75 mg of SHP647 SC injection every 4 weeks for an additional 72 weeks in the anterolateral right/left thigh or the deltoid area or the abdomen.
- Total: Total of all reporting groups
Arm/Group | SHP647 75 mg | SHP647 225 mg | Total
Number analyzed (Participants) | 164 | 166 | 330
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.5 (12.75) | 41.1 (13.68) | 40.8 (13.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 70 | 132
  Male | 102 | 96 | 198
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 160 | 160 | 320
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian | 11 | 15 | 26
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: Black or African American | 3 | 2 | 5
  Race: White | 148 | 143 | 291
  Race: More than one race | 0 | 0 | 0
  Race: Other | 2 | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Treatment-Emergent Serious Adverse Events (TESAEs), and Who Withdrew From Treatment Due to Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical investigation participant who was administered a product or medical device; the event did not need to necessarily have a causal relationship with the treatment or usage. A serious adverse event (SAE) was any untoward medical occurrence at any dose that resulted in death, was life threatening (immediate risk of death), required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, resulted in congenital anomaly/birth defect. Number of participants with TEAEs, STEAEs, and those withdrew from treatment due to TEAEs were reported.
Time Frame: From start of study drug administration up to 168 weeks
Population: SAS consisted of all enrolled participants who had received at least 1 dose of SHP647.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP647 75 mg | SHP647 225 mg
Number analyzed (Participants) | 164 | 166
Participants
  Participants with any TEAE | 146 | 147
  Participants with any TESAE | 34 | 40
  Participants who withdrew treatment due to TEAE | 12 | 23

2. Secondary Outcome: Percentage of Participants With Mucosal Healing at Week 16
Description: Mucosal healing was defined as an absolute Mayo subscore for endoscopy of 0 or 1 (based on centrally read score) as assessed by flexible sigmoidoscopy or colonoscopy. The Mayo score is a tool designed to measure disease activity for ulcerative colitis (UC). The Mayo scoring system ranges from 0 to 12 points and consists of 4 subscores (stool frequency, rectal bleeding, findings on flexible sigmoidoscopy, and physician's global assessment [PGA]) each graded 0 to 3 with the higher score indicating more severe disease activity. The percentage of participants with mucosal healing at week 16 was reported.
Time Frame: Week 16
Population: SAS consisted of all enrolled participants who had received at least 1 dose of SHP647.
Measure: Number; unit: Percentage of participants
Arm/Group | SHP647 75 mg | SHP647 225 mg
Number analyzed (Participants) | 164 | 166
Percentage of participants | 27.4 | 29.5

3. Secondary Outcome: Serum Trough Concentrations of SHP647 Versus Time
Description: Serum trough concentrations of SHP647 versus time was reported.
Time Frame: Baseline, Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72 and 156
Population: The pharmacokinetic (PK) set consisted of all participants who received at least 1 dose of SHP647 and for whom at least 1 postdose PK sample was collected. Here 'Number of Participants Analyzed' refers to the number of participants evaluable for specific timepoint.
Measure: Mean (Standard Deviation); unit: Micrograms/liter (ug/L)
Arm/Group | SHP647 75 mg | SHP647 225 mg
Number analyzed (Participants) | 163 | 164
Micrograms/liter (ug/L)
  Baseline: number analyzed (Participants) | 113 | 117
  Baseline | 6398.62 (8584.412) | 8064.41 (10629.768)
  Week 4: number analyzed (Participants) | 156 | 160
  Week 4 | 5496.56 (4026.759) | 16787.31 (7807.292)
  Week 8: number analyzed (Participants) | 155 | 157
  Week 8 | 6245.79 (3371.708) | 20345.29 (9286.956)
  Week 12: number analyzed (Participants) | 157 | 155
  Week 12 | 9038.72 (5540.836) | 23915.87 (10434.073)
  Week 16: number analyzed (Participants) | 141 | 149
  Week 16 | 10445.24 (6387.004) | 24772.35 (11970.153)
  Week 20: number analyzed (Participants) | 124 | 124
  Week 20 | 10928.76 (7900.859) | 25582.98 (11767.775)
  Week 24: number analyzed (Participants) | 115 | 123
  Week 24 | 11145.54 (8019.864) | 27832.20 (12469.086)
  Week 28: number analyzed (Participants) | 111 | 121
  Week 28 | 12978.11 (8772.285) | 27797.77 (13070.361)
  Week 32: number analyzed (Participants) | 110 | 119
  Week 32 | 12926.04 (8798.671) | 28381.93 (11748.573)
  Week 36: number analyzed (Participants) | 110 | 110
  Week 36 | 12785.55 (9182.501) | 29666.64 (13997.231)
  Week 40: number analyzed (Participants) | 102 | 109
  Week 40 | 13004.90 (9544.675) | 28947.34 (12151.971)
  Week 44: number analyzed (Participants) | 100 | 102
  Week 44 | 13337.50 (8620.549) | 29855.69 (13605.897)
  Week 48: number analyzed (Participants) | 104 | 99
  Week 48 | 14061.44 (9257.991) | 30010.61 (14014.183)
  Week 52: number analyzed (Participants) | 99 | 98
  Week 52 | 14192.83 (9326.176) | 28917.76 (14545.617)
  Week 56: number analyzed (Participants) | 98 | 97
  Week 56 | 15179.77 (10405.996) | 29985.88 (14122.172)
  Week 60: number analyzed (Participants) | 96 | 90
  Week 60 | 15133.54 (9673.602) | 29086.78 (12606.888)
  Week 64: number analyzed (Participants) | 91 | 91
  Week 64 | 15354.29 (10112.098) | 31613.08 (13712.478)
  Week 68: number analyzed (Participants) | 89 | 96
  Week 68 | 15584.38 (10407.781) | 30609.08 (14331.857)
  Week 72: number analyzed (Participants) | 88 | 90
  Week 72 | 15006.48 (9390.020) | 31342.89 (14012.311)
  Week 156: number analyzed (Participants) | 79 | 81
  Week 156 | 983.49 (1485.708) | 1893.88 (4530.680)

4. Secondary Outcome: Number of Participants With Positive Anti-drug (SHP647) Antibodies (ADA)
Description: The anti-drug antibodies (ADA) positive was defined as ADA log base 2 titer greater than or equal to (>=) 4.64. The number of participants with positive ADA was reported.
Time Frame: Baseline, Week 8, 16, 24, 40, 48, 64 and 156
Population: The SAS consisted of all enrolled participants who had received at least 1 dose of SHP647. Here, "number of participants analyzed" refers to the number of participants evaluable for this outcome at specific time points.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP647 75 mg | SHP647 225 mg
Number analyzed (Participants) | 164 | 166
Participants
  Baseline: number analyzed (Participants) | 148 | 153
  Baseline | 9 | 10
  Week 8: number analyzed (Participants) | 143 | 151
  Week 8 | 3 | 1
  Week 16: number analyzed (Participants) | 140 | 144
  Week 16 | 1 | 1
  Week 24: number analyzed (Participants) | 106 | 119
  Week 24 | 1 | 1
  Week 40: number analyzed (Participants) | 94 | 104
  Week 40 | 1 | 2
  Week 48: number analyzed (Participants) | 97 | 92
  Week 48 | 1 | 0
  Week 64: number analyzed (Participants) | 83 | 86
  Week 64 | 1 | 0
  Week 156: number analyzed (Participants) | 73 | 81
  Week 156 | 0 | 1

5. Secondary Outcome: Number of Participants With Positive Neutralizing Antibodies (NAb)
Description: The positive Neutralizing Antibodies (NAb) was defined as NAb titer greater than or equal to (>=) 0.903. The number of participants with NAb was reported. Here "inconclusive" refers to participants who were neither reported as positive nor negative for NAb and anti-drug antibodies (ADA) positive was defined as ADA log base 2 titer greater than or equal to (>=) 4.64.
Time Frame: Baseline, Week 8, 16, 24, 40, 48, 64 and 156
Population: Here, "number of participants analyzed" refers to the number of participants evaluable for this outcome at specific time points with non-missing ADA sample.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP647 75 mg | SHP647 225 mg
Number analyzed (Participants) | 148 | 153
Participants
  Baseline: Without +ADA | 139 | 143
  Baseline: With +ADA, with +NAb | 0 | 4
  Baseline: With +ADA, without +NAb | 0 | 1
  Baseline: With +ADA, with inconclusive NAb | 8 | 5
  Baseline: With +ADA, missing NAb | 1 | 0
  Week 8: Without +ADA: number analyzed (Participants) | 143 | 151
  Week 8: Without +ADA | 140 | 150
  Week 8: With +ADA, with +NAb: number analyzed (Participants) | 143 | 151
  Week 8: With +ADA, with +NAb | 1 | 1
  Week 8: With +ADA, without +NAb: number analyzed (Participants) | 143 | 151
  Week 8: With +ADA, without +NAb | 2 | 0
  Week 16: Without +ADA: number analyzed (Participants) | 140 | 144
  Week 16: Without +ADA | 139 | 143
  Week 16: With +ADA, with +NAb: number analyzed (Participants) | 140 | 144
  Week 16: With +ADA, with +NAb | 0 | 1
  Week 16: With +ADA, without +NAb: number analyzed (Participants) | 140 | 144
  Week 16: With +ADA, without +NAb | 1 | 0
  Week 24: Without +ADA: number analyzed (Participants) | 106 | 119
  Week 24: Without +ADA | 105 | 118
  Week 24: With +ADA, with +NAb: number analyzed (Participants) | 106 | 119
  Week 24: With +ADA, with +NAb | 0 | 1
  Week 24: With +ADA, without +NAb: number analyzed (Participants) | 106 | 119
  Week 24: With +ADA, without +NAb | 1 | 0
  Week 40: Without +ADA: number analyzed (Participants) | 94 | 104
  Week 40: Without +ADA | 93 | 102
  Week 40: With +ADA, with +NAb: number analyzed (Participants) | 94 | 104
  Week 40: With +ADA, with +NAb | 1 | 2
  Week 40: With +ADA, without +NAb: number analyzed (Participants) | 94 | 104
  Week 40: With +ADA, without +NAb | 0 | 0
  Week 48: Without +ADA: number analyzed (Participants) | 97 | 92
  Week 48: Without +ADA | 96 | 92
  Week 48: With +ADA, with +NAb: number analyzed (Participants) | 97 | 92
  Week 48: With +ADA, with +NAb | 1 | 0
  Week 48: With +ADA, without +NAb: number analyzed (Participants) | 97 | 92
  Week 48: With +ADA, without +NAb | 0 | 0
  Week 64: Without +ADA: number analyzed (Participants) | 83 | 86
  Week 64: Without +ADA | 82 | 86
  Week 64: With +ADA, with +NAb: number analyzed (Participants) | 83 | 86
  Week 64: With +ADA, with +NAb | 0 | 0
  Week 64: With +ADA, without +NAb: number analyzed (Participants) | 83 | 86
  Week 64: With +ADA, without +NAb | 1 | 0
  Week 156: Without +ADA: number analyzed (Participants) | 73 | 81
  Week 156: Without +ADA | 73 | 80
  Week 156: With +ADA, with +NAb: number analyzed (Participants) | 73 | 81
  Week 156: With +ADA, with +NAb | 0 | 0
  Week 156: With +ADA, without +NAb: number analyzed (Participants) | 73 | 81
  Week 156: With +ADA, without +NAb | 0 | 1

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to 168 weeks
Arm/Group | SHP647 75 mg | SHP647 225 mg
All-Cause Mortality (participants affected / at risk) | 1/164 | 0/166
Serious Adverse Events (participants affected / at risk) | 34/164 | 40/166
Other Adverse Events (participants affected / at risk) | 116/164 | 119/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SHP647 75 mg (N=164) | SHP647 225 mg (N=166)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Serous cystadenocarcinoma ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 15 (19) | 18 (19)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Non-Cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Arrhythmogenic right ventricular dysplasia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Serum sickness (Immune system disorders) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Meningitis listeria (Infections and infestations) | 0 (0) | 1 (1)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0)
Pelvic abscess (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Anastomotic fistula (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Blood iron decreased (Investigations) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Basilar migraine (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Typical aura without headache (Nervous system disorders) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SHP647 75 mg (N=164) | SHP647 225 mg (N=166)
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 (41) | 29 (42)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (15) | 18 (20)
Abdominal pain (Gastrointestinal disorders) | 9 (14) | 20 (33)
Colitis ulcerative (Gastrointestinal disorders) | 41 (52) | 36 (50)
Diarrhoea (Gastrointestinal disorders) | 11 (13) | 7 (11)
Nausea (Gastrointestinal disorders) | 8 (10) | 19 (20)
Vomiting (Gastrointestinal disorders) | 10 (10) | 7 (7)
Influenza like illness (General disorders) | 8 (11) | 9 (10)
Pyrexia (General disorders) | 14 (20) | 7 (10)
Bronchitis (Infections and infestations) | 10 (12) | 8 (12)
Clostridium difficile infection (Infections and infestations) | 11 (12) | 4 (4)
Gastroenteritis (Infections and infestations) | 18 (25) | 13 (17)
Influenza (Infections and infestations) | 8 (9) | 15 (19)
Nasopharyngitis (Infections and infestations) | 20 (27) | 28 (44)
Pharyngitis (Infections and infestations) | 2 (2) | 17 (20)
Sinusitis (Infections and infestations) | 7 (11) | 10 (14)
Upper respiratory tract infection (Infections and infestations) | 23 (34) | 20 (35)
Urinary tract infection (Infections and infestations) | 11 (15) | 10 (12)
Headache (Nervous system disorders) | 17 (23) | 21 (56)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (20) | 11 (12)
Rash (Skin and subcutaneous tissue disorders) | 8 (9) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2016-11-14): https://cdn.clinicaltrials.gov/large-docs/09/NCT01771809/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-02): https://cdn.clinicaltrials.gov/large-docs/09/NCT01771809/SAP_001.pdf